CLINICAL TRIAL: NCT03790462
Title: Evaluation of the Effect of Select Indian Ragas on Electrophysiological Parameters and Salivary Stress Markers - a Randomized Control Trial
Brief Title: Select Indian Ragas on Electrophysiological Parameters
Acronym: RAGA-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MS Ramaiah Medical College & Hospitals (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, KIRTHANA KUNIKULLAYA U, Principal Investigator, MS Ramaiah Medical College & Hospitals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2017-0174
Record Dates: First submitted 2018-12-26; First posted 2018-12-31 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Psychology, Social; Stress; Stress, Psychological
Keywords: Stress, Electroencephalogram,Indian Music, Electrocardiogram
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: It is a triple blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Music intervention group 1 (Experimental): Raga "A" will be played for 10 minutes & data collected.
  Interventions: Other: Music intervention
- Music intervention group 2 (Experimental): Raga "B" will be played for 10 minutes & data collected.
  Interventions: Other: Music intervention
- Music intervention group 3 (Experimental): Raga "C" will be played for 10 minutes & data collected.
  Interventions: Other: Music intervention
- Control group (No Intervention): Subject relaxes without music for 10 minutes and electrophysiological parameters will be collected

INTERVENTIONS:
Other: Music intervention — A raga out of 3 select Indian classical ragas "Puriya/Hindol/Todi" will be played for 10 minutes & data collected.
  Arms: Music intervention group 1; Music intervention group 2; Music intervention group 3

SUMMARY:
In India, music is predominantly used as entertainment. Despite ample vedic literature available on the beneficial effects of ragas in Indian music on human mind and body, scientific evidence for the same is extremely meager. This initial systematic study of 6 ragas, is an attempt to provide scientific evidence and validate the use of Indian classical music & thus present the scientific community with a new complementary therapy / non- pharmacological mode of treatment which could be used in prevention of various non-communicable diseases. In our previous study on prehypertensives and hypertensives, blood pressure (BP) reduced significantly after listening to Indian music [raga 'bhimpalas' (raga that normalizes BP)], daily for 3 months. Heart rate variability (HRV) recorded once on recruitment and end of study failed to show any change. On retrospection, we realised that the effect of only a single raga had been tested and the acute effects had not been elucidated. Specifically, EEG waves & cognitive ERPs were not studied. Hence a study encompassing all the 6 ragas that are known to normalize BP as given in literatures such as Gandharva Veda (Sama Veda) & Raga Chikitsa was planned. Among these, 3 ragas are now being studied & data analysis is in line. This proposal is to study the immediate electrophysiological changes with remaining 3 ragas. Music can be prescribed as a cheap and effective adjuvant in the treatment of hypertension along with other lifestyle modifications. To the best of our knowledge, there is scanty literature testing Indian ragas. Thus there is a great need to address this issue.

DETAILED DESCRIPTION:
INDIAN MUSIC: 'Raga' (musical scale) is a set of musical notes presented in an orderly manner in order to generate a melody out of the same. Matanga (9-10th century AD) in his work 'Brihaddeshi' was the earliest to define raga as "raga is that kind of sound composition consisting of melodic movements which has the effect of colouring the hearts of men". However, there have been very few studies which have used Indian classical music as an intervention for studying their health benefits. Gandharvaveda, a part of Sama veda, has mentioned various ragas to have myriad health benefits.Dr. Burnell has mentioned a manuscript named raga chikistsa in the collections of Saraswati Mahal Library in Tanjore which deals with the various ragas that can be used for curing various ailments. For example raga Malkauns is said to help in curing hypotension. Insomnic patients are said to benefit by usage of raga Behag. 'Heart Rate Variability' has become the conventionally accepted term to describe beat-to-beat alteration in HR, and RR intervals in ECG. The cause of HRV is considered to be respiratory sinus arrhythmia as well as low-frequency oscillations (0.1 Hz) associated with Traube-Hering-Mayer waves of BP . It was found that a decrease in HRV was a strong predictor of mortality after acute myocardial infarction . HRV is assessed by either time or frequency domain methods. EFFECT OF MUSIC ON BLOOD PRESSURE:Many studies have shown that there is a modification of cardiorespiratory parameters on repeated rhythymic recitation of a prayer, poetry or yoga mantra . So it is not surprising that music (rhythmic repetition of notes and tones) can also have similar effects. A number of studies have reported that listening to sedative music (slow tempo, legato phrasing, and minimal dynamic contrasts) can lead to decreased HR and BP. BP was shown to be proportional to the crescendo present in music, where as music with uniform emphasis reduced the BP .

Passive listening to music on a daily basis helped in reducing BP of 12 elderly subjects. The experimental group listened to selected songs for 25 minutes every day, for four weeks. BP was measured twice a week. There was a significant decrease in the mean BP: 11.8 mmHg in the SBP and 4.7 mmHg in the DBP . Elderly subjects have shown statistically significant reduction in SBP and DBP after 12-minute audio relaxation program . STUDIES ON EFFECT OF MUSIC ON HRV: Whether music causes an increase or decrease in HR, remains a mystery . Several studies reported that under various conditions music decreases sympathetic nervous system (SNS) and increases parasympathetic nervous system (PNS) activity as measured by HR and HRV, indicating physiological relaxation . No difference in HR or HRV was observed by a few investigators . However, an increase in HR has also been reported by some . SALIVARY STRESS MARKERS: The salivary glands receive sympathetic and parasympathetic innervations. The major enzyme that is released on sympathetic stimulation is alpha (α) amylase. Thus it is presumed that, changes in salivary alpha amylase indicate the activity of the SM system during stress. Further, both salivary cortisol and alpha amylase have been used by number of researchers recently to quantify stress or as biomarkers of stress. Nevertheless, it has also been put forth that salivary amylase activity is an index of plasma norepinephrine levels under a variety of stressful conditions. STUDIES ON EFFECT OF MUSIC ON EEG: In one study where EEG was recorded after giving alpha music to about ten subjects, it was observed that increase in the maximum amplitudes of Alpha waves either after 6 minutes or after 12 minutes of alpha music. However, the maximum amplitude of beta waves showed a decline of up to 40% from the initial value. These results, namely, the increase in Alpha activity and decrease in Beta activity indicate that subjects experience 'relaxed alertness'.

Setting: Medical college and Tertiary care hospital Case group (totally 3 groups) = 35 subjects in each group; a total sample of 105 Control group = 35 subjects Basis for sample size:Based on the study conducted by Okada et al, it was found that RMSSD (root mean square standard deviation of NN intervals on ECG) was 17.4±7.2 ms and 24.1±15.5 ms before and after music therapy with an effect size of 0.59 and power of 90% and confidence interval of 95%, the minimum sample size required for the present study was estimated to be 32.

Methods and materials: The effect of at least 3 different Indian classical music ragas on the autonomic functions and brain waves of subjects will be studied. Healthy subjects will be recruited from M S Ramaiah Instituitions. Selection bias will be avoided by randomization using computer generated random numbers. All numbers generated will be kept in an opaque and sealed envelope. The envelope will be opened by the research assistant after the baseline assessment of each participant and assigned to each of the seven groups randomly, into all intervention and control categories. Each group will randomly be assigned to listen to a particular raga using block randomization. The control group, the seventh group, will not receive any raga, but HRV,BP, EEG and saliva will be recorded and collected. Literature given in Gandharva veda and raga chikitsa will be used to choose ragas which have varied health benefits especially on the cardiovascular system. The ragas which have been said to normalize the BP are ahir bhairav, bhimpalas, hindol, puriya, kausikanada and todi. Ahir Bhairav, Kausi Kanada & Bhimpalas will be used for the present study. Detailed methodology: The investigators will include a few questions inquiring the subjects' preference of type of music, previous experience with music instrumental or vocal training and note the same. A general health check up will be done for all subjects. The BMI, waist hip ratio and BP in sitting position measured twice after five minutes rest (Sphygmomanometry) in between will be noted. A stress questionnaire (State Trait Anxiety Inventory) will be administered prior to and after intervention to assess the baseline level of stress and the change in stress levels after music intervention.

Subjects will be made to lie supine and relax for ten minutes. EEG electrodes will be applied according to 10-20 system. A baseline EEG (Galileo NT) and ECG in lead II for 10 minutes (Power lab 15 T Labchart by AD instruments) will be recorded. Baseline digital measurement of BP will be done. Saliva for baseline stress markers (cortisol and amylase) will be collected. All the subjects will be instructed to breathe at a rate of 6 breaths per minute, throughout the procedure that will be monitored by the software. After this, a raga from Indian classical music will be played for 10 minutes duration via earplugs connected to the laptop, during which time the recording of ECG and EEG will continue. The time of start of music will be marked using an event marker in the software. Post ten minutes, the music will be stopped and BP will be recorded and saliva will be collected. ECG and EEG recording will continue for another ten minutes to study any residual effects of music on the heart after which BP will be recorded and saliva will be collected again (end of 30 minutes procedure). Stress questionnaire will be administered at the end of the procedure. For those in control group baseline BP, ECG and EEG will be recorded for ten minutes under resting conditions. Saliva will be collected and stored. EEG will be analyzed using Galileo NT software. HRV will be analyzed using the software provided. The saliva samples will be centrifuged at 3000 rpm for 15 minutes and supernatant saliva stored at -20° C until further analysis for cortisol and amylase (ELISA).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Age group of 18-30 years
* Either gender will be included as autonomic functions change with age
* Non smokers
* Non alcoholics.

Exclusion Criteria:

* Any cardiovascular disorders,
* Renal disorders,
* Respiratory disorders,
* Endocrine disorders,
* Neurological problems
* Pregnancy,
* Body mass index (BMI)>30 kg/m2,
* Hearing problems,
* Psychiatric disorder
* Drugs which are known to affect the BP or autonomic status of the individual
* Other impairments that prevent the subject from performing few experimental procedures will be excluded.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 166 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-09 (Actual)

PRIMARY OUTCOMES:
Change in Blood pressure | Baseline, 10 minutes after music intervention & 10 minutes post intervention
  in mm Hg
Change in Electroencephalogram amplitude | Baseline, 10 minutes during music intervention & 10 minutes post intervention
  Change in Electroencephalogram (EEG) waves amplitude (in mV)
Change in Electroencephalogram Frequency | Baseline, 10 minutes during music intervention & 10 minutes post intervention
  Change in Electroencephalogram Frequency (in Hz)
Change in Stress using state trait anxiety inventory | Baseline, after 10 minutes of music intervention & 10 minutes post intervention
  State trait anxiety inventory score in numbers - It comprises separate self-report scales for measuring two distinct anxiety concepts: state anxiety and trait anxiety. The STAI-T scale consists of 20 statements that ask people to describe how they generally feel. The STAI-S scale also consists of 20 statements. Each question is rated on a 4-point scale (not at all, somewhat, moderately so, very much so). The range of possible scores for form Y of the STAI varies from a minimum score of 20 to a maximum score of 80 on both the STAI-T and STAI-S subscales. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).

SECONDARY OUTCOMES:
Change in Heart rate variability | Baseline, 10 minutes during music intervention & 10 minutes post intervention
  Analyzed in lead II of Electrocardiogram - time and frequency domain
Change in Salivary Cortisol | Baseline, after 10 minutes of music intervention & 10 minutes post intervention
  Change in level of salivary cortisol will be analyzed
Change in Salivary alpha amylase | Baseline, after 10 minutes of music intervention & 10 minutes post intervention
  Change in level of salivary alpha amylase will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: MEDHA RAO Y, MD, Study Chair — M S Ramaiah Medical college and hospitals
Locations (1):
- M S Ramaiah Medical college and hospitals, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No
Publications (Pre-press) may be shared with other researchers